CLINICAL TRIAL: NCT02318264
Title: Influence of Elastic Tape on Activation of the Quadriceps Muscle During Selected Resisted and Weight Bearing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Michelle Dolphin, Clinical Assistant Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SUMU-PT-KTAP1
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Results first posted 2022-05-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects; Changes Based on Duration of Tape Application; Direction of Kinesio Tape Application
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Distal to Proximal Tape (Experimental): Quadriceps muscle taped (Using Kinesio Tape) starting distal by knee and ending proximal by hip.
  Interventions: Device: Kinesio Tape
- Proximal to Distal Tape (Experimental): Quadriceps muscle taped (Using Kinesio Tape) starting proximal by hip and ending distal by knee.
  Interventions: Device: Kinesio Tape

INTERVENTIONS:
Device: Kinesio Tape — Elastic tape placed over the skin

SUMMARY:
This cross over design study will be used to determine the influence of elastic kinesiology tape on the speed and amplitude of quadriceps activation (anterior thigh) during selected resisted and weight bearing exercises.

DETAILED DESCRIPTION:
Objective: This cross over design study will be used to determine the influence of elastic kinesiology tape on the speed and amplitude of quadriceps activation (anterior thigh) during selected resisted and weight bearing exercises.

Background: Compliant tape, such as KiniseoⓇ Tape (KT), is highly elastic and claimed by the manufacturer to mimic skin. It is commonly used by physical therapists and sports medicine practitioners to treat musculoskeletal conditions and to enhance physical performance. The creators of KT teach a variety of applications techniques to affect the underlying musculature. Current theory regarding elastic tape application suggests that if the tape is applied over a muscle from the proximal to distal attachments, it will facilitate the underlying muscle while applying the tape from distal to proximal will inhibit the musculature.1 While studies have investigated the effect of elastic tape on muscle activation, few studies to date have compared the direction of application on muscle activation.2-7

Methods and Measures: Healthy subjects between 18-35 years old will be recruited from the Upstate Medical University community via email and word of mouth. Potential participants will report to the Institute for Human Performance and will be asked to complete all documentation including informed consent and a health-screening questionnaire. If eligible, qualified participants will perform 2 functional jumping exercises (vertical jump and single-leg triple hop for distance) 8 and isokinetic knee flexion and extension at 60 degrees/sec and 120 degrees/sec using the Biodex System 3 Pro Dynamometer (Biodex Medical Systems, Shirley, NY). The Biodex isokinetic machine has been shown to be a reliable and valid source of measuring peak torque, position and velocity.9 Surface electromyography (EMG) recordings will be collected from the vastus medialis and vastus lateralis during isokinetic testing. Testing will occur over four sessions. In the first session, baseline measurements and measurements immediately after KT application will be collected. In the second session, the participant will be retested after wearing the KT for up to two days (48 hours). This process will be repeated one week later during sessions three and four with KT applied in the opposite direction of the initial testing condition. KT application direction and the order of activities will be randomized for each participant.

ELIGIBILITY:
Eligible participants were between the ages of 18 to 35 and naïve to the use of kinesiology tape. Exclusion criteria included musculoskeletal injury to the lower extremities (within the previous year), past surgery to the lower extremities, or known allergy to adhesive tape.

All participants were screened for physical activity and exercise testing using the Physical Activity and Readiness Questionnaire (PAR-Q)15 (British Columbia Ministry of Health, British Columbia/Canada), resting vital signs, and American College of Sports Medicine guidelines for exercise testing. The Physical Activity and Readiness Questionnaire (PAR-Q)(British Columbia Ministry of Health) will be used as a general screen of exercise safety. Additionally, researchers will ask participants to identify possible cardiovascular and/or orthopedic risks to resistance exercise, dominant leg injuries/surgeries, and regarding history or familiarity of elastic tape. Subjects who are at risk due to recent (within the last year) musculoskeletal injury to lower extremities will be excluded from the study. Additionally, we will exclude subjects who report significant respiratory-cardiovascular disease, subjects with a history of surgery on their dominant leg, or individuals who have been trained in elastic tape theory and application. Any participant with a known allergy to adhesives will also be excluded from the study. Blood pressure and heart rate will be measured at the start of each session. Per ACSM's guidelines for exercise testing, if a participant's resting systolic blood pressure is greater than >200 mm Hg or diastolic BP is >110 mm Hg then he/she will be excluded from exercise testing and the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dolphin, DPT, Principal Investigator — SUNY Upstate Medical

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.

REFERENCES:
- [Result] Dolphin M, Brooks G, Calancie B, Rufa A. Does the Direction of Kinesiology Tape Application Influence Muscle Activation in Asymptomatic Individuals? Int J Sports Phys Ther. 2021 Feb 1;16(1):135-144. doi: 10.26603/001c.18799. PMID 33604143

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a crossover design. There were 15 subjects in total.
Groups:
- Distal to Proximal Tape, Then Proximal to Distal: Participants first received Quadriceps muscle taping (Using Kinesio Tape) starting distal by knee and ending proximal by hip, after a one week washout period, received quadriceps muscle taping starting proximal and ending distal.
  Kinesio Tape: Elastic tape placed over the skin
- Proximal to Distal Tape, Then Distal to Proximal: Participants first received quadriceps muscle taping (Using Kinesio Tape) starting proximal by hip and ending distal by knee, then after a one week washout period, received quadriceps muscle taping starting distal and ending proximal.
  Kinesio Tape: Elastic tape placed over the skin
Period: Overall Study
Arm/Group | Distal to Proximal Tape, Then Proximal to Distal | Proximal to Distal Tape, Then Distal to Proximal
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Distal to Proximal Tape, Then Proximal to Distal: Quadriceps muscle taped (Using Kinesio Tape) starting distal by knee and ending proximal by hip.
  Kinesio Tape: Elastic tape placed over the skin
- Proximal to Distal Tape, Then Distal to Proximal: Quadriceps muscle taped (Using Kinesio Tape) starting proximal by hip and ending distal by knee.
  Kinesio Tape: Elastic tape placed over the skin
- Total: Total of all reporting groups
Arm/Group | Distal to Proximal Tape, Then Proximal to Distal | Proximal to Distal Tape, Then Distal to Proximal | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (1.8) | 23.3 (1.8) | 23.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — This was by self report of sex.
  Participants
    Female | 5 | 5 | 10
    Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15
Hop Distance [Mean (Standard Deviation); unit: Centimeter] | 472.3 (88.1) | 468.4 (90.8) | 468.4 (90.8)
Vertical Jump Height [Mean (Standard Deviation); unit: centimeters] | 40.9 (18.5) | 41.6 (18.0) | 41.6 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: Vertical Jump Height Immediately Post Tape Administration
Description: Vertical Jump Height Immediately Post Tape Administration
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Distal to Proximal Tape: Quadriceps muscle taped (Using Kinesio Tape) starting distal by knee and ending proximal
  Kinesio Tape: Elastic tape placed over the skin
- Proximal to Distal Tape: Quadriceps muscle taped (Using Kinesio Tape) starting proximal by hip and ending distal.
  Kinesio Tape: Elastic tape placed over the skin
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
centimeters | 41.6 (18.3) | 41.1 (16.8)

2. Primary Outcome: Unilateral Three Hop for Distance Immediately Post Tape Administration
Description: Unilateral three hop for distance immediately post tape administration
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Distal to Proximal Tape: Quadriceps muscle taped (Using Kinesio Tape) starting distal by knee and ending proximal.
  Kinesio Tape: Elastic tape placed over the skin
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
centimeters | 471.5 (91.6) | 482.0 (99.5)

3. Secondary Outcome: EMG During Isokinetic Testing at 120 Degrees/Sec Immediately Post Tape Application
Description: EMG data were collected during the isokinetic testing at 120 degrees/sec Immediately Post Tape Application
Time Frame: Immediate
Measure: Mean (95% Confidence Interval); unit: Millivolts
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
Millivolts | .0052 [-.0058 to .0161] | -.0099 [-.0241 to .0043]

4. Secondary Outcome: EMG During Isokinetic Testing at 60 Degrees/Sec Immediately Post Tape Application
Description: EMG during isokinetic testing at 60 degrees/second Immediately Post Tape Application
Time Frame: Immediate
Measure: Mean (95% Confidence Interval); unit: Millivolts
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
Millivolts | .0053 [-.0074 to .0180] | -.0004 [-.0152 to .0145]

5. Secondary Outcome: Isokinetic Torque at 120 Degrees/Sec Immediately Post Tape Administration
Description: Isokinetic Torque at 120 Degrees/Second Immediately Post Tape Administration
Time Frame: Immediate
Measure: Mean (95% Confidence Interval); unit: Newton-Meters
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
Newton-Meters | 3.5 [-5.7 to 12.8] | 3.5 [-4.6 to 11.5]

6. Secondary Outcome: Isokinetic Torque at 60 Degrees/Sec Immediately Post Tape Administration
Description: Isokinetic Torque at 60 Degrees/Second Immediately Post Tape Administration
Time Frame: Immediate
Measure: Mean (95% Confidence Interval); unit: Newton-Meters
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
Number analyzed (Participants) | 15 | 15
Newton-Meters | 2.9 [-17.3 to 13.0] | -6.0 [-13.6 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during testing (1-2 hours per participant) but there was no followup. Participants were evaluated during testing.
Arm/Group | Distal to Proximal Tape | Proximal to Distal Tape
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
This was a small homogeneous sample of convenience with limited generalizability as the participants were young healthy adults without musculoskeletal injury. The study may be underpowered due to a small sample size of 15.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No